CLINICAL TRIAL: NCT04918654
Title: Automatic Sound Management 3.0 in a Single-unit Audio Processor
Acronym: RND3
Status: Completed | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: RND3_MED-EL_CRD_2020_03
Record Dates: First submitted 2021-05-31; First posted 2021-06-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Subjects

SUMMARY:
Cochlear implants are routine treatment for people with severe hearing loss. This study tests the RONDO 3, MED-EL's newest single-unit audio processor which comes with new features (Beamformer, Wind-Noise reduction, Ambient noise reduction, Transient noise reduction, Adaptive intelligence).

DETAILED DESCRIPTION:
MED-EL Cochlear Implants (CI) provide auditory sensations via electrical stimulation of the auditory pathways for severely to profoundly hearing-impaired individuals who obtain little or no benefit from acoustic amplification in the best aided condition. Front-end processing of acoustic signals picked up by the audio processor is routinely applied to provide optimal hearing performance under varying listening conditions. Automatic Sound Management (ASM) was introduced by MED-EL with the TEMPO+ audio processor and provided advanced compression and automatic gain management. With the SONNET audio processor, MED-EL introduced ASM 2.0, which added wind noise reduction and microphone directionality to the front-end processing. With the SONNET 2 audio processor, ASM 3.0 was implemented and the features ambient noise reduction, transient noise reduction and an adaptive intelligence (AI) were added. The RONDO 3 implements now ASM 3.0.

This study investigates the impact of ASM 3.0 as implemented in the RONDO 3 on CI users' speech performance and their subjective quality of hearing.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 18 years old
* Experienced user of a RONDO 3 (≥ 3 months) for the ear to be tested
* Post-lingual onset of severe to profound sensory-neural hearing loss on the ear to be tested
* A minimum of 40% speech recognition in the Freiburg Monosyllables Test in quiet at 65 dB SPL for the ear to be tested (at the last time tested in clinical routine)
* Signed and dated Informed Consent Form (ICF) before the start of any study-specific procedure.

Exclusion criteria

* Lack of compliance with any inclusion criteria
* CI user with contralateral hearing equal to or better than 30 dB (pure-tone average over the following frequencies: 250, 500, 1000, and 2000 Hz)
* Implanted with C40X, or C40C on the ear to be tested
* Implanted with an Auditory Brainstem Implant (ABI) or split electrode array
* Known allergic reactions to components of the investigational medical device (RONDO 3) or the SONNET 2
* Anything that, in the opinion of the Investigator, would (a) place the subject at increased risk, (b) preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post-lingually deafened adult cochlear implant users with a MED-EL device.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Speech in noise | Baseline
  Oldenburg Sentence Test in noise (S0 N±90 N180)

SECONDARY OUTCOMES:
Quality of Hearing | Baseline
  Hearing Implant Sound Quality Index (HISQUI). Min score: 16, Max score 133. Higher scores mean a better outcome.
Device Satisfaction | Baseline
  Audio Processor Satisfaction Questionnaire. Min score: 0, Max score 10. Higher scores mean a better outcome.
User Satisfaction | Baseline
  Product-specific questionnaire. The questionnaire is not reporting a single score on a scale (min/max score not applicable).
Speech in noise | Baseline
  Oldenburg Sentence Test in noise (S0 N±90 N180)
Speech in noise | Baseline
  Oldenburg Sentence Test in noise (S0 N0)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Büchner, Prof. Dr., Principal Investigator — Hals-Nasen-Ohrenklinik der Medizinischen Hochschule Hannover
Locations (1):
- MHH - Medizinische Hochschule Hannover, Hanover, Germany

REFERENCES:
- [Result] Buchner A, Rottmann T, Lenarz T, Lesinski-Schiedat A, Aschbacher E, Fruhauf F, Bracker T, Billinger-Finke M. Clinical improvement of speech perception in noise with Automatic Sound Management 3.0. Hear Res. 2025 Dec;468:109445. doi: 10.1016/j.heares.2025.109445. Epub 2025 Oct 4. PMID 41115327